CLINICAL TRIAL: NCT04343417
Title: Biorepository to Support Research in Kidney Diseases
Status: Enrolling by invitation | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000027890; 1K23DK117065-01A1 (NIH); R01DK128087 (NIH)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Acute Interstitial Nephritis; Kidney Diseases
Keywords: Kidney; Kidney Disease; Acute Kidney Injury; Kidney biopsy; Kidney Biorepository
MeSH Terms: conditions — Acute Kidney Injury; Acute Tubulointerstitial Nephritis; Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood (serum, plasma, and DNA extraction), urine samples, kidney tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biorepository: Participants who contributed biospecimen samples (kidney tissue, blood, urine, DNA).

SUMMARY:
To support advances in the understanding of pathophysiology and therapies of kidney diseases by creating a BioBank of kidney tissue, DNA, plasma, and urine from patients with kidney diseases.

DETAILED DESCRIPTION:
A biorepository of human samples to support research to advance understanding of human kidney diseases will be created. Clinically, kidney diseases are detected by blood and urine laboratory tests. However, the underlying cause of kidney disease is often not clear on blood and urine tests. In such cases, a clinician may choose to perform a kidney biopsy to establish the diagnosis. Patients who are scheduled to undergo a kidney biopsy will be invited to participate in this proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a clinically indicated kidney biopsy
* English or Spanish speaking

Exclusion Criteria:

* Under 18 years or age
* Known pregnancy
* Additional vulnerable individuals (incarcerated, institutionalized, or otherwise unable to participate in the study)
* Inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The biorepository is a prospective cohort study of subjects with kidney diseases, who are scheduled to undergo a kidney biopsy at Yale New Haven Hospital (York St. or St. Raphael's campus) as part of the routine clinical care and agree to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2035-08-01 (Estimated)

PRIMARY OUTCOMES:
Histological diagnosis | 5 years
  Histological diagnosis of kidney disease determined by evaluation by renal pathologists

SECONDARY OUTCOMES:
Occurrence of chronic kidney disease, end stage kidney disease or death | 10 years
  Track outcomes in participants recruited for up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G Moledina, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, York Street Campus, New Haven, Connecticut
  - Yale New Haven Hospital Saint Raphael Campus, New Haven, Connecticut